CLINICAL TRIAL: NCT04788108
Title: Oral Progesterone for Prevention of Miscarriage in Threatened Abortion: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Oral Progesterone for Prevention of Miscarriage in Threatened Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Head of Placental Related Diseases Research Unit, Principal Investigator, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 177/2021
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Threatened Abortion
Keywords: threatened abortion
MeSH Terms: conditions — Abortion, Threatened | interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dydrogesterone (Active Comparator): dydrogesterone 10 mg by mouth every 12 hours until 1 week after bleeding stops or until 6 weeks.
  Interventions: Drug: Dydrogesterone
- Placebo (Placebo Comparator): placebo by mouth every 12 hours until 1 week after bleeding stops or until 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dydrogesterone — Dydrogesterone tablet
  Arms: Dydrogesterone
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
This study evaluates the effectiveness of oral dydrogesterone in preventing miscarriage in threatened abortion. Half of participants will receive oral dydrogesterone, while the other half will receive oral placebo.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy with gestational age 6 - 20 weeks
* threatened abortion
* confirmed intrauterine pregnancy with a viable fetus by ultrasound

Exclusion Criteria:

* history of recurrent miscarriage
* having endocervical polyp
* having infection such as pneumonia, pyelonephritis, septicemia
* having autoimmune diseases such as systemic lupus erythematosus, systemic sclerosis, rheumatoid arthritis
* having cancer
* having coagulation defect
* allergy to dydrogesterone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
continue pregnancy more than 20 weeks gestation | at 20 weeks gestation
  percentage of cases with continue pregnancy more than 20 weeks gestation

SECONDARY OUTCOMES:
preterm delivery less than 34 weeks | at 34 weeks gestation
  percentage of delivery less than 34 weeks
preterm delivery less than 37 weeks | at 37 weeks gestation
  percentage of delivery less than 37 weeks
placenta previa | 31 weeks
  percentage of placenta previa
abruptio placenta | 31 weeks
  percentage of abruptio placenta
Intrauterine growth restriction | 31 weeks
  percentage of intrauterine growth restriction
neonatal complications | 31 weeks
  percentage of newborn with respiratory distress syndrome, intraventricular hemorrhage, necrotizing enterocolitis, death
side effects | 6 weeks
  percentage of side effects such as headache, nausea/vomiting
compliance | 6 weeks
  percentage of complete drug use
maternal satisfaction | 6 weeks
  percentage of good satisfaction
time until bleeding stops | 6 weeks
  time from first bleeding until bleeding stops

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University, Faculty of Medicine, Department of Obstetrics and Gynecology
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Gynecology. ACOG Practice Bulletin No. 200: Early Pregnancy Loss. Obstet Gynecol. 2018 Nov;132(5):e197-e207. doi: 10.1097/AOG.0000000000002899. PMID 30157093
- [Background] Mirza FG, Patki A, Pexman-Fieth C. Dydrogesterone use in early pregnancy. Gynecol Endocrinol. 2016;32(2):97-106. doi: 10.3109/09513590.2015.1121982. Epub 2016 Jan 22. PMID 26800266
- [Background] Schindler AE, Campagnoli C, Druckmann R, Huber J, Pasqualini JR, Schweppe KW, Thijssen JH. Classification and pharmacology of progestins. Maturitas. 2003 Dec 10;46 Suppl 1:S7-S16. doi: 10.1016/j.maturitas.2003.09.014. PMID 14670641
- [Result] Omar MH, Mashita MK, Lim PS, Jamil MA. Dydrogesterone in threatened abortion: pregnancy outcome. J Steroid Biochem Mol Biol. 2005 Dec;97(5):421-5. doi: 10.1016/j.jsbmb.2005.08.013. Epub 2005 Nov 15. PMID 16293412
- [Result] Pandian RU. Dydrogesterone in threatened miscarriage: a Malaysian experience. Maturitas. 2009 Dec;65 Suppl 1:S47-50. doi: 10.1016/j.maturitas.2009.11.016. Epub 2009 Dec 14. PMID 20005647
- [Result] El-Zibdeh MY, Yousef LT. Dydrogesterone support in threatened miscarriage. Maturitas. 2009 Dec;65 Suppl 1:S43-6. doi: 10.1016/j.maturitas.2009.11.013. Epub 2009 Dec 14. PMID 20007011